CLINICAL TRIAL: NCT06854588
Title: Point-of-care Ultrasound Screening of Thoracic Aortic Aneurysm in Hypertensive Patients in the Emergency Department
Brief Title: POCUS Screening for TAA in Hypertensive Patients in the ED
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Colin Graham, Professor, Chinese University of Hong Kong
Other Study IDs: NTEC-2024-753
Record Dates: First submitted 2025-02-12; First posted 2025-03-03 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Thoracic Aortic Aneurysm (TAA); Aortic Dissection
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hypertensive patients presenting to the emergency department: 1. Adult patients aged ≥ 18 years attending the ED during the study period
  2. Known history of hypertension or newly diagnosed hypertension in the ED
  Interventions: Diagnostic Test: Point-of-care ultrasound

INTERVENTIONS:
Diagnostic Test: Point-of-care ultrasound — POCUS screening will be conducted to measure the maximum diameters at end diastole of the aortic root, ascending aorta, aortic arch, and descending thoracic aorta.

SUMMARY:
The investigators are going to recruit hypertensive patients in the emergency department of Prince of Wales Hospital. Point-of-care ultrasound of the aorta and measurements of the aortic diameter will be obtained. Other relevant clinical data will also be obtained for analysis. The primary outcome is the number of patients with a maximum aortic diameter of ≥ 4.5 cm and/or ≥ 50% localized enlarged diameter relative to the adjacent normal segment as indicated by POCUS.

DETAILED DESCRIPTION:
Investigators trained with point-of-care ultrasound (POCUS) will recruit hypertensive patients in the emergency department (ED) of Prince of Wales Hospital. POCUS will be performed using a handheld ultrasound device to visualise the aortic root, ascending aorta, aortic arch and descending aorta. Measurements of the diameter will be obtained from different segments of the thoracic aorta for analysis. The definition of aortic aneurysm is a maximum aortic diameter of ≥ 4.5 cm and/or ≥ 50% localized enlarged diameter relative to the adjacent normal segment as indicated by POCUS. The primary outcome is the prevalence of thoracic aortic aneurysm (TAA) in hypertensive patients in the ED. The secondary outcomes include the number of patients with confirmed TAA as verified by CTA, BMI for all participants, the number of CTA scans conducted for TAA confirmation, the number of surgical interventions performed among TAA patients, the ICU admission rate, ICU length of stay, hospital length of stay and mortality, proportion of adequate visualisation of POCUS studies obtained, agreement of aortic diameter measurement between CTA and POCUS, and signs and symptoms of TAA patients presenting to the ED. In addition, the investigators will assess the 28-day all-cause mortality and any advanced imaging done outside the ED.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥ 18 years attending the ED during the study period
* Known history of hypertension or newly diagnosed hypertension in the ED

Exclusion Criteria:

* Known history of aortic aneurysm or dissection
* Previous thoracic aortic interventions or endovascular stenting
* Patients in cardiopulmonary resuscitation
* Traumatic patients
* Patients refuse to participate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: hypertensives patients attending the emergency department without known history of aortic diseases.
Sampling Method: Non-Probability Sample
Enrollment: 1483 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
number of patients with a dilated aorta | Day 1
  is the number of patients with a maximum aortic diameter of ≥ 4.5 cm and/or ≥ 50% localized enlarged diameter relative to the adjacent normal segment as indicated by POCUS

SECONDARY OUTCOMES:
number of patients with confirmed TAA | through study completion, an average of 1 year
  number of patients with confirmed TAA as verified by CTA

OTHER OUTCOMES:
BMI for all participants | at the time of recruitment
  BMI in kg/m^2
number of CTA scans | through study completion, an average of 1 year
  number of CTA scans conducted for TAA confirmation
number of surgical interventions | from recruitment to 28 days after
  number of surgical interventions performed among TAA patients
ICU and hospital length of stay | through study completion, an average of 1 year
  ICU and hospital length of stay among patients with treatment for TAA
mortality | from recruitment to 28 days after
  28-day mortality in both TAA and non-TAA patients
proportion of adequate visualisation of POCUS studies obtained | up to 1 year
  proportion of adequate visualisation of POCUS studies (%) obtained during the recruitment period
agreement of aortic diameter measurement | from recruitment to 28 days after if CTA is performed
  agreement of aortic diameter measurement between CTA and POCUS in cm

CONTACTS AND LOCATIONS:
Overall Officials: Colin A Graham, Professor, Principal Investigator — Accident and Emergency Medicine Academic Unit, CUHK
Locations (1):
- Prince of Wales Hospital, Shatin, NT, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Not allowed by the ethics committee